CLINICAL TRIAL: NCT03013712
Title: A Clinical Research of CAR T Cells Targeting EpCAM Positive Cancer
Acronym: CARTEPC
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Chengdu Medical College (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CARTEPC-001
Record Dates: First submitted 2017-01-03; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Colon Cancer; Esophageal Carcinoma; Pancreatic Cancer; Prostate Cancer; Gastric Cancer; Hepatic Carcinoma
MeSH Terms: conditions — Colonic Neoplasms; Esophageal Neoplasms; Pancreatic Neoplasms; Prostatic Neoplasms; Stomach Neoplasms; Carcinoma, Hepatocellular | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CAR-T cell immunotherapy (Experimental): Enrolled patients will receive CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at EpCAM antigen by infusion.
  Interventions: Biological: CAR-T cell immunotherapy

INTERVENTIONS:
Biological: CAR-T cell immunotherapy — This CAR-T cell immunotherapy with a novel specific Chimeric antigen receptor aiming at EpCAM antigen.

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of EpCAM-specific CAR T Cells infusion for EpCAM positive Cancer.

DETAILED DESCRIPTION:
This study is being conducted to evaluate the safety and efficacy of Chimeric antigen receptor (CAR) T cells targeting EpCAM in treating patients with EpCAM positive cancer. In the research, the investigators design a novel CAR consists of a EpCAM targeting antibody scFv with two intracellular signaling domains derived from CD3 zeta and CD28. Autologous T cells will be gene-engineered with the CAR gene using a lentivirus vector. Prior to T cell infusion, the patients will be subjected to preconditioning treatment. The infusion dose is (1-10)×106 EpCAM-CAR positive T cells/kg, and the specific cells numbers depends on the situation of individual CAR-T cells preparation. The way of infusion is vascular interventional mediated or endoscopy, and the cells perfusion process would lasts 15min to 30min, and the specific time depends on patent's tumor-burdened state. After T cell infusion, the patients will be evaluated for 24 months for adverse reactions, persistence of CAR T cells and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory EpCAM positive cancer.
2. KPS > 60.
3. Life expectancy>3 months.
4. Gender unlimited, age from 18 years to 80 years.
5. Assessable lesions with a minimum size of 10mm by CT scan or MRI.
6. Acceptable organ function Hematology:

   * Absolute neutrophil count greater than 800/mm^3 without the support of filgrastim.
   * White blood cell (WBC) (> 2000/mm^3).
   * Platelet count greater than 50,000/mm^3.
   * Hemoglobin greater than 9.0 g/dl.
7. No other serious diseases(autoimmune disease, immunodeficiency etc.).
8. Adequate cardiac function (LVEF ≥ 40%).
9. No other tumors.
10. Patients volunteer to participate in the research.

Exclusion Criteria:

1. Allergic to cytokines.
2. Uncontrolled active infection.
3. Acute or chronic GVHD.
4. MODS.
5. Treated with T cell inhibitor.
6. HIV affected.
7. Pregnancy.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-01; Primary Completion 2018-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Toxicity profile of the EpCAM targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0 | up to 24 months
  Observe and handle the toxicity profile of the EpCAM targeted CAR T cells with Common Toxicity Criteria for Adverse Effects (CTCAE) version 4.0

SECONDARY OUTCOMES:
Survival time of anti-EpCAM CAR T cells in vivo | up to 24 months
  Detect the existence of CAR-T cells in the blood of participants through flow cytometry
Anti-tumor efficacy of CAR-T therapy by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1 | up to 24 months
  Anti-tumor efficacy of CAR-T therapy for patients with EpCAM positive cancers was assessed by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-an Li, PhD, Study Chair — First Affiliated Hospital of Chengdu Medical College
Locations (1):
- IEC of Chengdu Medical College, Chendu, China

IPD SHARING:
Plan to Share IPD: No